CLINICAL TRIAL: NCT05525533
Title: Supporting Young Women's Reproductive Health by Harnessing Prosociality Among Drug Shopkeepers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study is linked to a parent study. The parent study was stopped prematurely; as a result this study was also stopped prematurely.
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Berkeley (Other); Health for a Prosperous Nation (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: R03HD109561-01 (NIH); R03HD109561-01 (NIH)
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Results first posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Hiv; Contraception
Keywords: Drug shops; Pro-sociality; Adolescent health; HIV self-testing; Contraception
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial; the investigators will phase in the 2 interventions (Private and Public Feedback) on a staggered basis. All shops will receive No Feedback during the first 6 months. One third of shops (~N=40) will be assigned to No Feedback between 6-12 months; one third of shops (~N=40) will be assigned to Private Feedback between 6-12 months; one third of shops (~N=40) will be assigned to Public Feedback between 6-12 months.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No feedback (Experimental): AGYW customer feedback will be collected but not shared with shopkeepers
  Interventions: Behavioral: Harnessing prosocial and social image motivations for behavior change
- Private feedback (Experimental): Biweekly summarized reports of AGYW customer feedback will be given directly to shopkeepers
  Interventions: Behavioral: Harnessing prosocial and social image motivations for behavior change
- Public feedback (Experimental): Shopkeepers will get biweekly summarized reports of AGYW customer feedback, gold stars reflecting the level of AGYW customer feedback (e.g., 1-5 star rating) will be placed in the shop in a visible location, and shopkeepers will be invited to an awards ceremony every 6 months to recognize shopkeepers who receive high levels of positive AGYW customer feedback
  Interventions: Behavioral: Harnessing prosocial and social image motivations for behavior change

INTERVENTIONS:
Behavioral: Harnessing prosocial and social image motivations for behavior change — The investigators will collect AGYW customer feedback using a short USSD-based survey and randomize whether shopkeepers receive 1) No feedback; 2) Private feedback; or 3) Public feedback

SUMMARY:
The goal of the study is to operationalize and test the preliminary impact of providing regular customer feedback from adolescent girls and young women (AGYW) to drug shopkeepers on the distribution of contraceptives and HIV self-testing to AGYW over 12 months.

DETAILED DESCRIPTION:
The investigators will cross-randomize 120 drug shops enrolled in the parent Malkia Klabu effectiveness cluster-randomized controlled trial (CRCT; NCT05357144), stratified by CRCT study arm, to one of three initial conditions: 1. No feedback. AGYW customer feedback will be collected, but not shared with the shopkeeper. 2. Private feedback. Biweekly summarized reports of AGYW customer feedback will be given directly to shopkeepers. 3. Public feedback: Shopkeepers will get biweekly summarized reports of AGYW customer feedback, gold stars reflecting the level of AGYW customer feedback (e.g., 1-5 star rating) will be placed in the shop in a visible location, and shopkeepers will be invited to an awards ceremony every 6 months to recognize shopkeepers who receive high levels of positive AGYW customer feedback. The investigators will phase in the 2 interventions (Private and Public Feedback) on a staggered basis to control for both shop-specific and time-specific trends for the primary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Shopkeepers enrolled in the parent CRCT

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenny X Liu, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- Tanzania (2):
  - Mwanza Province, Mwanza
  - Shinyanga, Shinyanga

IPD SHARING:
Plan to Share IPD: Yes
The investigators will make the data and associated documentation available to users upon request and only under a data-sharing agreement with the study team that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying the data after analyses are completed.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The SP, SAP, and ICF will be made available on the Open Science Framework (OSF) within 12 months recruitment.
  Study results will be posted to OSF and Clinical Trials within 12 months of completion of data collection.
Access Criteria: Everything posted to OSF and Clinical Trials will be made publicly available.

REFERENCES:
- [Background] Hunter LA, McCoy SI, Rao A, Mnyippembe A, Hassan K, Njau P, Mfaume R, Liu JX. Designing drug shops for young women in Tanzania: applying human-centred design to facilitate access to HIV self-testing and contraception. Health Policy Plan. 2021 Nov 11;36(10):1562-1573. doi: 10.1093/heapol/czab084. PMID 34313728
- [Background] Chiu C, Hunter LA, McCoy SI, Mfaume R, Njau P, Liu JX. Sales and pricing decisions for HIV self-test kits among local drug shops in Tanzania: a prospective cohort study. BMC Health Serv Res. 2021 May 6;21(1):434. doi: 10.1186/s12913-021-06432-1. PMID 33957903
- [Derived] Chiu C, Mnyippembe A, Sheira LA, Packel L, Katabaro E, Maokola W, Liu JX. Boosting health provider performance with non-financial incentives: A cluster-randomized controlled trial in Tanzania. PLoS One. 2025 Sep 11;20(9):e0330989. doi: 10.1371/journal.pone.0330989. eCollection 2025. PMID 40934247

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Please note that for the purposes of this study, "participants" refer to each drug shop owner or representative enrolled in the study. Each drug shop enrolled one participant. There are no other participants in this study. Shops were recruited on a rolling basis within each arm. The wards are geographical units that were the unit of randomization (cluster). All shops within each ward had the same treatment assignment.
Units Other Than Participants: Ward
Groups:
- No Feedback: Participants will receive no feedback for 12 months.
  No feedback: AGYW customer feedback will be collected but not shared with shopkeepers
  Harnessing prosocial and social image motivations for behavior change: The investigators will collect AGYW customer feedback using a short USSD-based survey and randomize whether shopkeepers receive 1) No feedback; 2) Private feedback; or 3) Public feedback
- No Feedback (Phase 1) - Private Feedback (Phase 2): Participants will receive no feedback for 6 months and then private feedback for 6 months.
  Private feedback: Biweekly summarized reports of AGYW customer feedback will be given directly to shopkeepers
  Harnessing prosocial and social image motivations for behavior change: The investigators will collect AGYW customer feedback using a short USSD-based survey and randomize whether shopkeepers receive 1) No feedback; 2) Private feedback; or 3) Public feedback
- No Feedback (Phase 1) - Public Feedback (Phase 2): Participants will receive no feedback for 6 months, then public feedback for 6 months.
  Public feedback: Shopkeepers will get biweekly summarized reports of AGYW customer feedback, gold stars reflecting the level of AGYW customer feedback (e.g., 1-5 star rating) will be placed in the shop in a visible location, and shopkeepers will be invited to an awards ceremony every 6 months to recognize shopkeepers who receive high levels of positive AGYW customer feedback
  Harnessing prosocial and social image motivations for behavior change: The investigators will collect AGYW customer feedback using a short USSD-based survey and randomize whether shopkeepers receive 1) No feedback; 2) Private feedback; or 3) Public feedback
Period: Phase 1 - No Feedback
Arm/Group | No Feedback | No Feedback (Phase 1) - Private Feedback (Phase 2) | No Feedback (Phase 1) - Public Feedback (Phase 2)
Started | 44; 12 Ward | 49; 15 Ward | 51; 14 Ward
Completed | 44; 12 Ward | 49; 15 Ward | 51; 14 Ward
Not Completed | 0; 0 Ward | 0; 0 Ward | 0; 0 Ward
Period: Phase 2 - No, Private or Public Feedback
Arm/Group | No Feedback | No Feedback (Phase 1) - Private Feedback (Phase 2) | No Feedback (Phase 1) - Public Feedback (Phase 2)
Started | 44; 12 Ward | 49; 15 Ward | 51; 14 Ward
Completed | 44; 12 Ward | 49; 15 Ward | 51; 14 Ward
Not Completed | 0; 0 Ward | 0; 0 Ward | 0; 0 Ward

BASELINE CHARACTERISTICS:
Groups:
- No Feedback: No feedback for 12 months.
  No feedback: AGYW customer feedback will be collected but not shared with shopkeepers
  Harnessing prosocial and social image motivations for behavior change: The investigators will collect AGYW customer feedback using a short USSD-based survey and randomize whether shopkeepers receive 1) No feedback; 2) Private feedback; or 3) Public feedback
- No Feedback - Private Feedback: No feedback for 6 months, private feedback for 6 months.
  Private feedback: Biweekly summarized reports of AGYW customer feedback will be given directly to shopkeepers
  Harnessing prosocial and social image motivations for behavior change: The investigators will collect AGYW customer feedback using a short USSD-based survey and randomize whether shopkeepers receive 1) No feedback; 2) Private feedback; or 3) Public feedback
- No Feedback - Public Feedback: No feedback for 6 months, public feedback for 6 months.
  Public feedback: Shopkeepers will get biweekly summarized reports of AGYW customer feedback, gold stars reflecting the level of AGYW customer feedback (e.g., 1-5 star rating) will be placed in the shop in a visible location, and shopkeepers will be invited to an awards ceremony every 6 months to recognize shopkeepers who receive high levels of positive AGYW customer feedback
  Harnessing prosocial and social image motivations for behavior change: The investigators will collect AGYW customer feedback using a short USSD-based survey and randomize whether shopkeepers receive 1) No feedback; 2) Private feedback; or 3) Public feedback
- Total: Total of all reporting groups
Arm/Group | No Feedback | No Feedback - Private Feedback | No Feedback - Public Feedback | Total
Number analyzed (Participants) | 44 | 49 | 51 | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (10.6) | 38.6 (14.5) | 30.2 (8.7) | 34.4 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex unknown for 2 participants
  Participants
    number analyzed (Participants) | 44 | 47 | 51 | 142
    Female | 26 | 32 | 32 | 90
    Male | 18 | 15 | 19 | 52
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Quantity of HIV Self-test Kits Distributed
Description: Mean number of HIV self-test kits sold per shop every month
Time Frame: 12 months
Population: It was pre-specified to report this outcome measure at the 12-month time point after all participants received this sequence of interventions.
Measure: Mean (Standard Deviation); unit: Items sold
Arm/Group | No Feedback | Private Feedback | Public Feedback
Number analyzed (Participants) | 44 | 49 | 51
Items sold | 153.53 (203.84) | 181.13 (209.49) | 239.13 (286.70)
Statistical Analysis 1: Comparison: No Feedback vs Private Feedback; Test type: Superiority; Regression, Linear; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [-1.87 to 2.24]
Statistical Analysis 2: Comparison: No Feedback vs Public Feedback; Test type: Superiority; Regression, Linear; Mean Difference (Final Values) = 1.55, 95% CI 2-sided [-0.73 to 3.82]

2. Primary Outcome: Quantity of HIV Self-test Kits Distributed
Description: Mean number of HIV self-test kits distributed per shop every 2 weeks
Time Frame: 18 months
Population: The customer feedback intervention ended due to the early termination of the parent study. As a result, these data were not collected beyond 12 months, therefore we cannot report on this 18 month outcome. The 12-month outcome is reported under Outcome 1. This study used the same participants as as the parent study and when the parent study terminated so did this study. All data collection ceased when the parent study terminated, after 12 months of this study.
Arm/Group | No Feedback | Private Feedback | Public Feedback
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Quantity of Sexual and Reproductive Health Products Sold
Description: Mean number of sexual and reproductive health products sold per shop every month
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Items sold
Arm/Group | No Feedback | Private Feedback | Public Feedback
Number analyzed (Participants) | 44 | 49 | 51
Items sold | 9.68 (9.38) | 9.27 (9.06) | 10.70 (9.95)
Statistical Analysis 1: Comparison: No Feedback vs Private Feedback; Test type: Superiority; Regression, Linear; Mean Difference (Final Values) = 7.58, 95% CI 2-sided [-2.92 to 18]
Statistical Analysis 2: Comparison: No Feedback vs Public Feedback; Test type: Superiority; Regression, Linear; Mean Difference (Final Values) = 16, 95% CI 2-sided [0.64 to 31]

4. Primary Outcome: Quantity of Contraceptives Distributed
Description: Mean number of contraceptives distributed per shop every 2 weeks
Time Frame: 18 months
Population: The customer feedback intervention ended due to the early termination of the parent study. As a result, these data were not collected beyond 12 months, therefore we cannot report on this 18 month outcome. The 12-month outcome is reported under Outcome 3. This study used the same participants as as the parent study and when the parent study terminated so did this study. All data collection ceased when the parent study terminated, after 12 months of this study.
Arm/Group | No Feedback | Private Feedback | Public Feedback
Number analyzed (Participants) | 0 | 0 | 0

5. Primary Outcome: Quantity of All Products Sold
Description: Mean number of all products sold per shop per month
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: items sold
Arm/Group | No Feedback | Private Feedback | Public Feedback
Number analyzed (Participants) | 44 | 49 | 51
items sold | 11.87 (34.19) | 17.05 (36.14) | 20.11 (51.09)
Statistical Analysis 1: Comparison: No Feedback vs Private Feedback; Test type: Superiority; Regression, Linear; Mean Difference (Final Values) = 47, 95% CI 2-sided [-18 to 113]
Statistical Analysis 2: Comparison: No Feedback vs Public Feedback; Test type: Superiority; Regression, Linear; Mean Difference (Final Values) = 113, 95% CI 2-sided [38 to 189]

6. Secondary Outcome: Quantity of Condoms Sold
Description: Mean number of condoms sold per shop every month
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: items sold
Arm/Group | No Feedback | Private Feedback | Public Feedback
Number analyzed (Participants) | 44 | 49 | 51
items sold | 3.19 (11.16) | 6.36 (21.18) | 4.63 (11.12)
Statistical Analysis 1: Comparison: No Feedback vs Private Feedback; Test type: Superiority; Regression, Linear; Mean Difference (Final Values) = 3.63, 95% CI 2-sided [-1.37 to 8.63]
Statistical Analysis 2: Comparison: No Feedback vs Public Feedback; Test type: Superiority; Regression, Linear; Mean Difference (Final Values) = 1.50, 95% CI 2-sided [-1.50 to 4.50]

7. Secondary Outcome: Quantity of Emergency Contraception Sold
Description: Mean number of emergency contraception sold per shop every month
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: items sold
Arm/Group | No Feedback | Private Feedback | Public Feedback
Number analyzed (Participants) | 44 | 49 | 51
items sold | 1.56 (5.06) | 2.60 (6.57) | 3.28 (9.96)
Statistical Analysis 1: Comparison: No Feedback vs Private Feedback; Test type: Superiority; Regression, Linear; Mean Difference (Final Values) = 1.32, 95% CI 2-sided [-0.36 to 7.30]
Statistical Analysis 2: Comparison: No Feedback vs Public Feedback; Test type: Superiority; Regression, Linear; Mean Difference (Final Values) = 3.38, 95% CI 2-sided [-0.54 to 7.30]

8. Secondary Outcome: Quantity of Oral Contraception Sold
Description: Mean number of oral contraception sold per shop every month
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: items sold
Arm/Group | No Feedback | Private Feedback | Public Feedback
Number analyzed (Participants) | 44 | 49 | 51
items sold | 4.21 (13.83) | 3.30 (8.58) | 7.04 (19.98)
Statistical Analysis 1: Comparison: No Feedback vs Private Feedback; Test type: Superiority; Regression, Linear; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [-3.38 to 3.72]
Statistical Analysis 2: Comparison: No Feedback vs Public Feedback; Test type: Superiority; Regression, Linear; Mean Difference (Final Values) = 7.57, 95% CI 2-sided [0.42 to 15]

9. Secondary Outcome: Quantity of Pregnancy Tests Sold
Description: Mean number of pregnancy tests sold per shop every month
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: items sold
Arm/Group | No Feedback | Private Feedback | Public Feedback
Number analyzed (Participants) | 44 | 49 | 51
items sold | 2.91 (6.99) | 4.79 (8.79) | 5.15 (11.80)
Statistical Analysis 1: Comparison: No Feedback vs Public Feedback; Test type: Superiority; Regression, Linear; Mean Difference (Final Values) = 2.46, 95% CI 2-sided [-0.11 to 5.02]
Statistical Analysis 2: Comparison: No Feedback vs Public Feedback; Test type: Superiority; Regression, Linear; Mean Difference (Final Values) = 3.29, 95% CI 2-sided [0.33 to 6.25]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | No Feedback | Private Feedback | Public Feedback
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/49 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/49 | 0/51
Other Adverse Events (participants affected / at risk) | 0/44 | 0/49 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-19): https://cdn.clinicaltrials.gov/large-docs/33/NCT05525533/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-19): https://cdn.clinicaltrials.gov/large-docs/33/NCT05525533/ICF_001.pdf